CLINICAL TRIAL: NCT06162767
Title: A Randomized Controlled Study of Optimized Sweet Procedure Versus Ivor-Lewis Procedure Esophagectomy in Adenocarcinoma of Esophagogastric Junction
Brief Title: Cancer of Esophagogastric Junction: Optimized Sweet Versus Ivor-Lewis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-186-02
Record Dates: First submitted 2023-11-14; First posted 2023-12-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-06

CONDITIONS: Esophagogastric Junction Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivor-Lewis Procedure (Active Comparator): Arm A: Esophagectomy was conducted through right side thoracotomy plus midline laparotomy approach: Ivor-Lewis Procedure.
  Interventions: Procedure: Esophagectomy by Ivor-Lewis Procedure
- Optimized Sweet Procedure (Active Comparator): Arm B: Esophagectomy was conducted by single-incision thoracoscope combined with laparoscopy with the patient in a right oblique side position at 45 degrees: Optimized Sweet Procedure.
  Interventions: Procedure: Esophagectomy by Optimized Sweet Procedure

INTERVENTIONS:
Procedure: Esophagectomy by Ivor-Lewis Procedure — Esophagectomy was conducted by Ivor-Lewis Procedure.
  Arms: Ivor-Lewis Procedure
Procedure: Esophagectomy by Optimized Sweet Procedure — Esophagectomy was conducted by Optimized Sweet Procedure.
  Arms: Optimized Sweet Procedure

SUMMARY:
This study is being done to see whether Optimized Sweet Procedure is superior than the Ivor-Lewis Procedure Esophagectomy with better long-term outcome and acceptable postoperative short-term outcome or not.

DETAILED DESCRIPTION:
Esophagogastric junction carcinoma is a prevalent malignancy within the human digestive system, ranking as the sixth leading cause of cancer-related deaths worldwide. Current national and international guidelines advocate for a comprehensive approach primarily centered around surgical intervention for the management of esophagogastric junction carcinoma. This preference stems from the fact that lymph node metastasis in such patients can occur simultaneously in the abdominal region and the lower mediastinum. Consequently, conventional options like the Ivor Lewis and Sweet procedures are routinely recommended due to their capability to encompass tumor resection, margin clearance, and lymph node dissection. However, traditional Sweet procedures are associated with higher surgical trauma and increased postoperative complications. With the evolution of single-incision thoracoscopy, we have leveraged the advantages of minimally invasive techniques and innovatively devised an Optimized "totally thoracoscopic Sweet procedure".In this study, a randomized controlled trial will enroll 240 patients diagnosed with esophagogastric junction carcinoma to compare the therapeutic efficacy between the Optimized Sweet Procedure and the Ivor-Lewis Procedure. Postoperative follow-ups will be conducted to analyze pre-discharge indicators and five-year postoperative outcomes, examining the correlation between the two surgical procedures in terms of postoperative quality of life, mortality rates, and survival rates, aiming to explore whether the Optimized Sweet Procedure is superior to the Ivor-Lewis Procedure Esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative diagnosis confirmed by esophagogastroduodenoscopy showing an Esophagogastric junction mass, with histopathological confirmation of malignancy, specifically Siewert Type II;
2. Preoperative blood pressure controlled below 160/100 mmHg, blood glucose levels within 5.6 to 11.2 mmol/L, and normal functioning of major organs such as heart, lungs, liver, and kidneys. Main criteria include a Goldman cardiac risk index of grade 1 or 2; pulmonary function tests indicating predicted postoperative forced expiratory volume in 1 second (FEV1) > 40%, and carbon monoxide diffusion capacity (DLCO) ≥ 40%; total bilirubin < 1.5 times the upper limit of normal; Alanine amioTransferase (ALT) and Aspartate Transaminase (AST) < 2.5 times the upper limit of normal; creatinine ≤ 1.25 times the upper limit of normal and creatinine clearance ≥ 60 mL/min;
3. Enhanced thin-slice CT scan of the thorax and abdomen showing a tumor with a maximum diameter not exceeding 5 cm, and lymph nodes in the thorax and abdomen with a short diameter not exceeding 1 cm, clinically staged as CT1-2N0-1M0 (8th edition JACC staging);
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-1;
5. All relevant examinations completed within 14 days before surgery;
6. Patients capable of understanding the study and providing informed consent by signing the consent form.

Exclusion Criteria:

Patients who have undergone prior anti-tumor therapy (such as radiotherapy, chemotherapy, immunotherapy, etc.) before surgery; individuals with a history of other malignancies; patients presenting with secondary primary cancer at the time of enrollment; those with a history of prior unilateral thoracic or abdominal major surgeries; pregnant or lactating women; individuals with interstitial pneumonia, pulmonary fibrosis, or severe emphysema; uncontrolled infections; severe mental illness; and those with a history of severe heart disease, congestive heart failure, myocardial infarction, or angina attacks within the last six months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Postoperative morbidity | 3 years
Postoperative mortality | 3 years
locoregional recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Louqian Zhang, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China